CLINICAL TRIAL: NCT01605500
Title: Investigation of the Utility of the Audible Alert in Current Generation Medtronic ICDs
Brief Title: Utility of the Audible Alert in Current Generation Medtronic Implantable Cardioverter-defibrillators
Status: Completed | Type: Observational
Sponsor: Englewood Hospital and Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: E-12-445
Record Dates: First submitted 2012-05-18; First posted 2012-05-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Patients With a Generation 2 Medtronic Implantable Cardioverter-defibrillator(ICD)
Keywords: ICD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medtronic ICDs: Patients with Generation 2 Medtronic ICDs

SUMMARY:
The purpose of this study is to determine whether the alert tones emitted by the latest generation of Medtronic implantable cardioverter-defibrillators (ICDs) are audible to patients.

ICD patients can have difficulties hearing the beeps, which are designed to notify patients of possible lead or generator malfunction. In fact, the only published study of this issue, conducted at Englewood Hospital and Medical Center, revealed that only 50% of patients with older Medtronic devices were able to hear alerts. Since then, modifications to the alert have been made by Medtronic. This study will establish the "real-world" value of these changes and also provide useful in vivo information regarding the validity of the in vitro techniques which have been used thus far to design the Patient Alert feature.

DETAILED DESCRIPTION:
There will be a single study visit. In a quiet examination room, the Patient Alert tones will be demonstrated to the subjects. Subsequently, this will be repeated with a wall air conditioner turned on. The subjects will then be asked to complete a three-part questionnaire regarding their perceptions of the Patient Alert tones.

Data analysis will include overall ability to hear tones, as well as subgroup analysis according to gender, age, and BMI.

Simultaneously, in order to calculate the loudness of the alert tones, digital recordings will be obtained using two microphones located near the subject. These digital recordings will be analyzed, and a loudness value will be calculated. The loudness value is a calculated index, devised by Medtronic, which incorporates frequency and intensity. Data analysis will include a correlation between loudness value and patient characteristics, and between loudness value and ability of subjects to perceive the tones.

ELIGIBILITY:
Inclusion Criteria:

* Previous insertion of a Medtronic Generation 2 ICD (Consulta, Secura, Concerto II, Virtuoso II, Maximo II devices) not fewer than 7 days prior to study entry
* Able to provide informed consent

Exclusion Criteria:

* Known deafness
* Recent (fewer than 6 weeks) ICD pocket surgery
* Non-Generation 2 Medtronic ICD
* Pocket hematoma
* Pocket infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have a Generation 2 Medtronic implantable cardioverter-defibrillator (ICD)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Audibility | participants will be tested during a single, routine clinic visit - the average duration for each patient will be 30 minutes
  how frequently patients are able to detect the alert tones

SECONDARY OUTCOMES:
Loudness value | 1 month
  digital recordings of the tones will be analyzed to determine the loudness value
  loudness value is a calculated index, devised by Medtronic, which incorporates frequency and intensity

CONTACTS AND LOCATIONS:
Overall Officials: Grant Simons, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States

REFERENCES:
- [Background] Simons EC, Feigenblum DY, Nemirovsky D, Simons GR. Alert tones are frequently inaudible among patients with implantable cardioverter-defibrillators. Pacing Clin Electrophysiol. 2009 Oct;32(10):1272-5. doi: 10.1111/j.1540-8159.2009.02480.x. Epub 2009 Aug 18. PMID 19691679